CLINICAL TRIAL: NCT04390360
Title: Development and Evaluation of Smartphone App for Initiation of Protective Ventilation. Clinical Impact of Instrumental Dead Space Reduction on Physiologic Parameter Based on the Smartphone App
Brief Title: Smartphone Application for Initiation of Protective Ventilation. Clinical Impact of Instrumental Dead Space Reduction
Acronym: Ventilo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 21750
Record Dates: First submitted 2020-04-20; First posted 2020-05-15 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: ARDS, Human; Mechanical Ventilation Complication; Humidifier Lung
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Protective ventilation with HME (Other): Protective ventilation + HME
  Interventions: Procedure: Protective ventilation with HME
- Protective ventilation with Heated humidifier (Other): Protective ventilation + HH
  Interventions: Procedure: Protective ventilation with Heated humidifier
- Implementation of protective ventilation (Other): Protective ventilation implementation
  Interventions: Procedure: Protective ventilation implementation
- Tidal Volume reduction (Other): Tidal volume reduction
  Interventions: Procedure: Tidal Volume reduction

INTERVENTIONS:
Procedure: Protective ventilation implementation — In this condition, we will implement the protective ventilation related with gender and height . A blood gas will be performed at before protective ventilation implementation and at the end of this condition.Time condition 30 minutes
  Arms: Implementation of protective ventilation
Procedure: Protective ventilation with HME — In this condition, the patient will received protective ventilation with a Heat Moisture Exchanger (HME). A blood gas will be performed at the end of this condition.Time condition 30 minutes
  Arms: Protective ventilation with HME
Procedure: Protective ventilation with Heated humidifier — In this condition, the patient will received protective ventilation with a Heated humidifier. A blood gas will be performed at the end of this condition.Time condition 30 minutes
  Arms: Protective ventilation with Heated humidifier
Procedure: Tidal Volume reduction — n this condition, we will reduce Tidal volume (with smartphone application calculation) to obtain the same alveolar ventilation (PaCO2) obtained on the HME condition
  Arms: Tidal Volume reduction

SUMMARY:
Clinical evaluation of a new educative tools (Smartphone application) based on impact of instrumental dead space reduction after initiation of protective ventilation during mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Mechanical ventilation (control,assist control or SIMV mode)
* haemodynamic stability (vasopressor < 0.2 ug/kg/min)
* no prone position schedule in the next 2 hours following procedure inclusion
* presence of an Arterial catheter

Exclusion Criteria:

* ECMO or anticipate ECMO
* body temperature < 36.0 for post operative patient (cardiac surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
PaCO2 Variation | 60 minutes post intervention
  The primary outcome is to evaluate the PaCO2 variation at the end of condition 2 (after 30 minutes with protective ventilation+ HME) and condition 4 (30 minutes after Tidal volume reduction + Heater humidifier).
  Variation <= 10% of PaCO2
PaCO2 Variation | 120 minutes post intervention
  The primary outcome is to evaluate the PaCO2 variation at the end of condition 2 (after 30 minutes with protective ventilation+ HME) and condition 4 (30 minutes after Tidal volume reduction + Heater humidifier).
  Variation <= 10% of PaCO2

SECONDARY OUTCOMES:
Correlation between PCO2 variation and alveolar ventilation variation | 60 and 90 minutes post intervention
  We will compare PaCO2 level variation and the alveolar ventilation variation to establish correlation.
  Correlation variation under 10% will be significative
Hemodynamic impact vs pH | Baseline, 30, 60, 90 and 120 minutes post intervention
  Cardiac echographic measurement (LeftVentricularEjectionFraction) in relation with acidosis status
Hemodynamic impact vs pH | Baseline, 30, 60, 90 and 120 minutes post intervention
  Cardiac echographic measurement (RightVentricularEjectionFraction) in relation with acidosis status
Hemodynamic impact vs pH | Baseline, 30, 60, 90 and 120 minutes post intervention
  Cardiac echographic measurement Arterial pulmonary pressure) in relation with acidosis status

CONTACTS AND LOCATIONS:
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval, Québec, Canada